CLINICAL TRIAL: NCT04741711
Title: Impact of Ultrasound-guided Therapeutic Management of Ambulatory Patients With Heart Failure : An Open-label Randomized Clinical Trial
Brief Title: AMBulatory UltraSound for Heart Failure Management
Acronym: AMBUSH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Pr. Nicolas GIRERD, MD,PhD, Central Hospital, Nancy, France
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019PI094
Record Dates: First submitted 2021-01-29; First posted 2021-02-05 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group (Experimental): The heart failure treatments will be guided by the results of the lung ultrasound and the evaluation of the inferior vena cava
  Interventions: Procedure: An ultrasound (lung and inferior vena cava) will be performed and the heart failure treatments will be guided by the results of the lung ultrasound and the evaluation of the inferior vena cava.
- Control group (Other): Usual care (i.e. without ultrasound guidance) will be provided.
  Interventions: Procedure: Usual care without ultrasound guidance

INTERVENTIONS:
Procedure: An ultrasound (lung and inferior vena cava) will be performed and the heart failure treatments will be guided by the results of the lung ultrasound and the evaluation of the inferior vena cava. — An ultrasound (lung and inferior vena cava) will be performed and the heart failure treatments will be guided by the results of the lung ultrasound and the evaluation of the inferior vena cava. The choice of congestion treatment modalities to be implemented is left to the investigators' discretion, in accordance with European practice guidelines.
  Arms: Interventional group
Procedure: Usual care without ultrasound guidance — Usual care (i.e. without ultrasound guidance)
  Arms: Control group

SUMMARY:
AMBUSH study is a multicenter randomized, controlled, open-label clinical trial (PROBE (Prospective Randomized Open Blinded End-point) type).

The main objective of AMBUSH study is to assess the effect of therapeutic management guided by pulmonary ultrasound and the assessment of the inferior vena cava in patients with heart failure seen in an ambulatory (outpatient) setting on a mixed clinical-biological endpoint (including variations of natriuretic peptides - NtProBNP) at 30 days.

DETAILED DESCRIPTION:
Secondary objectives are:

A. To assess the effect of therapeutic management guided by pulmonary ultrasound and inferior vena cava assessment on the risk of cardiovascular death and hospitalization for heart failure at 30 days.

B. Describe the proportion of ultrasound congestion (pulmonary and inferior vena cava data) in patients free from clinical congestion at baseline in the intervention group and in all patients at D30 visit.

C. Evaluate the association of ultrasound congestion (pulmonary and inferior vena cava assessment) with serum concentrations of natriuretic peptides at baseline and D30 visit.

D. Evaluate the association of variations in ultrasound congestion (pulmonary and evaluation of the inferior vena cava) and variations in natriuretic peptides between baseline and D30 visit.

E. Compare the proportion of ultrasound and clinical congestion in patients in the intervention group and in the control group at baseline and on D30 visit.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 and over
* Heart failure (regardless of left ventricular ejection fraction)
* Diagnosis of heart failure established more than 3 months ago
* Absence of significant clinical signs of congestion on clinical examination (absence of crackles and lower limbs oedema greater than perimalleolar oedema)
* Affiliation to social security
* Receiving complete information about research organization and signed informed consent.

Exclusion Criteria:

* Natriuretic peptides result, carried out during the previous 30 days, available at the inclusion consultation
* Pulmonary or pleural pathology preventing reliable acquisition of lung ultrasound images: severe emphysema, chronic pleurisy, pulmonary fibrosis.
* Suspicion of cardiac amyloidosis or proven amyloidosis,
* Patient with severe primary heart valve disease
* Pregnant woman, parturient or nursing mother
* Adult person subject to a legal protection measure (guardianship, curatorship, safeguard of justice)
* Person deprived of liberty by a judicial or administrative decision,
* Person subject to psychiatric care pursuant to Articles L. 3212-1 and L. 3213-1 of the Public Health Code.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2027-06-15 (Estimated)

PRIMARY OUTCOMES:
Death within 30 days (composite endpoint) | Within 30 days
  The primary endpoint will rank patients from worst to most favourable outcome during the trial. It will be a hierarchical composite of events as described by Felker in 2010 (PMID 20841546).
Hospitalization for heart failure within 30 days (composite endpoint) | Within 30 days
  The primary endpoint will rank patients from worst to most favourable outcome during the trial. It will be a hierarchical composite of events as described by Felker in 2010 (PMID 20841546).
Changes in N-terminal pro b-type natriuretic peptide (NtProBNP) between randomization and D30 (composite endpoint) | Between randomization and Day 30
  The primary endpoint will rank patients from worst to most favourable outcome during the trial. It will be a hierarchical composite of events as described by Felker in 2010 (PMID 20841546).

SECONDARY OUTCOMES:
Cardiovascular death | Within 30 days
  Within the combined outcome of CV death or hospitalization for heart failure. Outcomes will be adjudicated blinded from randomization arm
Ultrasound pulmonary congestion defined ≥3 B-lines on two intercostal spaces bilaterally (8-point method) and systemic congestion defined as an inferior vena cava diameter 21 mm or greater and/or a low variation during the respiratory cycle | At baseline in the intervention group and in all patients at Day 30 post inclusion
Circulating levels of natriuretic peptides (NtProBNP) | At baseline and Day 30
Changes in natriuretic peptides (NtProBNP) | Between baseline and Day 30.
Ultrasound congestion defined as in B / and clinical congestion evaluated according to the EVEREST and ASCEND scores | At baseline in the intervention group and in all patients at the Day 30.

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - CHU de Besançon, Besançon
  - CH de Mulhouse, Mulhouse
  - CHRU de Reims, Reims
  - CHR de Metz, Thionville
  - CHRU de Nancy, Vandœuvre-lès-Nancy